Baptist Health IRB IRB approval: 8/25/2022 Last approval: 8/25/2022 Expires: 8/24/2023 IRB#: 21-152

General Consent for parent(s)/legal guardian(s)

**Title of the Study**: Promote Healthy Lifestyle Behaviors for Adolescents with Mental Health Conditions

Principal Investigator: Rachel Sharp, BSN, RN, CPN, DNP-FNP Student, Florida State

University College of Nursing

Faculty Advisor: Dr. Geneva Scott-King, DNP-MSN-FNP-C, Teaching Faculty II, Florida State

University College of Nursing

You are being invited to take part in a research study. Please find below information about this research for you to think about before you decide to take part. Ask us if you have any questions about this information or the research before you decide to take part.

## **Key Information for You to Consider**

**Statement of the Research Study.** You are being invited to volunteer to take part in our research study. It is up to you whether you choose to take part or not. There will be no penalty or loss of benefits to you if you choose not to take part or decide later not to take part.

**Purpose**. The reason that we are doing this research is to find out more about the impact of an educational intervention on improving healthy lifestyle behaviors (nutrition, physical activity, screen time, and sleep).

**Duration.** We think that taking part in our study will last one-month.

**Research Activities.** Within a two-week period, you will be asked to complete a pre-survey survey that takes approximately 10-15 minutes and attend an online Zoom educational session that takes approximately 45 minutes. One-month after completing the pre-survey and participating in educational session, you will be asked to take a post-intervention survey that will take approximately 10-15 minutes.

**Risks:** The risks or discomforts to you of taking part in this study include **minimal risk.** That means you may feel embarrassed with some of the questions that I will ask, or you may feel uncomfortable answering some of my questions. Taking the surveys and joining the educational presentation may make you tired. You will **NOT** be asked for your name during this study.

**Benefits:** As a result of taking part in this research, we think that you may improve healthy lifestyle behaviors of your child.

#### What is this study about?

Researchers at Florida State University are studying Best Practices to Promote Healthy Lifestyle Behaviors for Adolescents with a Mental Health Condition(s). Researchers are interested in finding out about the impact of an educational intervention on improving healthy lifestyle behaviors (nutrition, physical activity, screen time, and sleep) among adolescents (12-17 years old) and their parents/legal guardian(s). You are invited to take part in the study because you are the parent or legal guardian of an adolescent with a diagnosed mental health condition(s). You are one of 60 persons (30 adolescent-parent/legal guardian dyads) to take part in this study. Your involvement in the study is expected to last one-month.

Baptist Health IRB IRB approval: 8/25/2022 Last approval: 8/25/2022 Expires: 8/24/2023

IRB#: 21-152

# What will happen during this research?

If you agree to be in this research, your participation will include answering a pre-and post-intervention surveys regarding your knowledge and behaviors on healthy lifestyle behaviors and attending a 45-minute zoom educational session on healthy lifestyle knowledge and behaviors.

- You will receive a project pre-survey survey will be sent out the middle to end of September 2022. You will have 2 weeks to complete pre-survey and attend a zoom educational session.
- A reminder email will be sent to participants on to complete survey/educational video. The educational session will be recorded and sent via email 1 week after education session.
- Participants will then receive a post-survey 1 month after finishing survey/educational video middle to end of October 2022.
- Study will be completed by early November 2022.

We will tell you about any new information that may affect your willingness to continue to take part in this research.

# What will you do to protect my privacy?

The results of the study may be published or presented, but no information that may identify you will ever be provided or released in publications or presentations. We will take steps to protect your privacy and confidentiality. These steps include:

- You will **not** be asked to provide your name or the name of your adolescent during this study. You will be asked to provide your date of birth.
- Your pre- and post-intervention survey responses will be tracked via the email you provide in the survey.
- Only members of the study team will have access to the subjects' identifiable information.
- Information will be secured/encrypted when stored, at rest, used, analyzed or when transmitted through REDCap.
- You will not be asked to provide identifiable information/biospecimens during this study.
- Parents/Legal guardians will be required to complete the survey and provide adolescent assent prior to the survey being completed by the adolescent.

Despite taking steps to protect your privacy or the confidentiality of your identifiable information, we cannot guarantee that your privacy or confidentiality will be protected. For

Baptist Health IRB IRB approval: 8/25/2022 Last approval: 8/25/2022 Expires: 8/24/2023

IRB#: 21-152

example, if you tell us something that makes us believe that you or others have been or may be physically harmed, we may need to report that information to the appropriate agencies.

Individuals and organizations responsible for conducting or monitoring this research may be permitted access to and inspect the research records. This includes the Florida State University Institutional Review Board (FSU IRB) and Baptist Health Institutional Review Board (Baptist Health IRB), which reviewed this study.

The information collected as part of this research will not be used or distributed for future research studies, even if all of your identifiers are removed.

#### What are the risks of harms or discomforts associated with this research?

The risks of harms or discomforts associated with the research are that there is minimal risk associated with this study. That means you may feel embarrassed with some of the questions that I will ask, or you may feel uncomfortable answering some of my questions. Taking the survey and joining the educational presentation may make you tired.

# How might I benefit from this research?

Personal benefits you may get from this study are that you may improve healthy lifestyle behaviors.

### What is the compensation for the research?

If you agree to take part in this research study, each adolescent-parent/legal guardian dyad will be provided with a \$5.00 Amazon E-Gift Card for each completion of the 3 activities associated with the project: pre-survey, educational presentation, and post-survey. E-Gift Cards will be sent to email provided via survey (REDCap) for adolescent-parent/legal guardian dyad. You will receive compensation within 24-48hrs after completing each activity of the project. Total compensation for dyad is \$15.00 in Amazon E-Gift Cards when project is completed in its entirety. Withdrawing or discontinuing taking part in the study will preclude participants from earning further incentive.

# What will happen if I choose not to participate?

It is your choice to participate or not to participate in this research. Participation is voluntary.

#### Is my participation voluntary, and can I withdraw?

Taking part in this research study is your decision. Your participation in this study is voluntary. You do not have to take part in this study, but if you do, you can stop at any time. Your decision whether to participate will not affect your relationship with the project researchers or FSU. Withdrawing or discontinuing taking part in the study will preclude participants from earning any further incentive/compensation.

If you withdraw from the study, the data collected to the point of withdrawal will not be used and will be deleted.

Baptist Health IRB IRB approval: 8/25/2022 Last approval: 8/25/2022 Expires: 8/24/2023 IRB#: 21-152

# Can I be removed from the research without my OK?

We may remove you from the research study without your approval. Reasons we would do this include

- Non-legal guardians
- Females that are pregnant before or after the start of the study

## Who do I talk to if I have questions?

If you have questions, concerns, or have experienced a research-related injury, contact the research team at:

Mrs. Rachel Sharp, BSN, RN, CPN FSU DNP-FNP Student Florida State University College of Nursing rls14c@my.fsu.edu

Dr. Geneva Scott-King, DNP-MSN-FNP-C Teaching Faculty II Florida State University College of Nursing gscottking@fsu.edu

The Florida State University Institutional Review Board ("IRB") is overseeing this research. The FSU IRB is a group of people who perform official independent review of research studies before studies begin to ensure that the rights and welfare of participants are protected. If you have questions about your rights or wish to speak with someone other than the research team, you may contact:

Florida State University IRB 2010 Levy Drive, Suite 276 Tallahassee, Florida 32306 850-644-7900 humansubjects@fsu.edu

or

Baptist Health IRB 904-202-2127 Baptist.IRB@bmcjax.com

Baptist Health IRB IRB approval: 8/25/2022 Last approval: 8/25/2022 Expires: 8/24/2023 IRB#: 21-152